CLINICAL TRIAL: NCT05511129
Title: Tolerance and Efficacy of Amiklin Administration During Nosocomial Infections Complicating COVID-19 in the ICU
Acronym: ReaMax2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ReaMax2
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; Nosocomial Infection
MeSH Terms: conditions — COVID-19; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The most severe infectious episodes are managed in intensive care. Classically, a distinction is made between sepsis, an infection associated with an inappropriate, excessive response of the immune system, responsible for organ dysfunction, and septic shock, during which, within the potential dysfunctions, hemodynamic alteration is central, requiring the introduction of catecholamines. The seriousness of these disorders, particularly because of their potential short-term severity, requires immediate treatment. The treatment of severe infections is based on the control of microbial proliferation, particularly bacterial. In this context, the speed of antibiotic therapy is associated with patient prognosis. If the administration of antibiotic therapy is an emergency during severe infections, particularly in situations of septic shock, its choice is decisive in the effectiveness of management and in the prognosis of the patient. Prior to microbiological results, antibacterial treatment is probabilistic. In spite of these numerous parameters, failure of probabilistic antibiotic therapy, due to a spectrum unsuited to the pathogens, is described in 15 to 30% of cases. In order to limit the risk of inappropriate treatment, it is recommended that broad-spectrum antibiotic therapy be used in states of shock of infectious origin. Because of their bactericidal properties, their kinetics of effectiveness, their marked post-antibiotic effect, their bioavailability in the plasma sector, and their synergy with beta-lactams, aminoglycosides are often recommended in combination in the initial probabilistic treatment. Despite numerous studies and extensive international experience with aminoglycosides, their real value in the management of severe infections remains uncertain, leading to contradictory information depending on whether one is interested in their benefit in the treatment of identified infections or in the probabilistic treatment of severe conditions.

During the management of severe intensive care patients, the pharmacokinetics of drugs, especially antibiotics, are considerably modified. As a result, monitoring of plasma, or better, tissue concentrations of antibiotics is suggested by learned societies, although their practical realization is still very limited by numerous obstacles.

Misuse of aminoglycosides is associated with a risk of acute renal failure, centered on the tubular toxicity of the antibiotic. While the risks associated with inappropriate frequency of administration are currently modest, those associated with high peak concentration, responsible for an increase in the duration of renal exposure, are not well known.

COVID-19 is also associated with a high risk of impaired renal function. The effect of aminoglycoside administration in the context of COVID-19 remains unknown. Our goal is to determine whether the presence of COVID-19 associates with an elevated risk of renal failure when prescribing aminoglycoside.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age ≥ 18 years
* Hospitalization for respiratory Covid-19
* Patient hospitalized in the ICU or Respiratory Department for a PCR-confirmed respiratory infection with COVID-19
* French-speaking patient

Exclusion Criteria:

* Patient with a severe psychiatric disorder
* A dying patient
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his or her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with age ≥ 18 years, hospitalized for respiratory Covid-19 in the ICU or Respiratory Department for a PCR-confirmed respiratory infection with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changed risk of renal failure | Month 3
  This outcome corresponds to the evolution of renal function, calculated as the difference 1/ between the creatinine and urea values at entry and the maximum value and 2/ between the creatinine and urea values at entry and the value at discharge.

SECONDARY OUTCOMES:
Effect of maximum serum concentration of Amikacin on renal function | Month 3
  This outcome corresponds to the percentage of patients with return to normal creatinine and urea values.
Effect of Amikacin administration on the probability of recovery of renal function | Month 3
  This outcome corresponds to the number of days between the maximum creatinine and urea value and normalization of the values. A "normal" value at discharge is defined as a value less than 1.25 times the entry value.
Effect of Amikacin administration on the rate of recovery of renal function | Month 3
  This outcome corresponds to the percentage of deaths during the resuscitation stay.

CONTACTS AND LOCATIONS:
Overall Officials: François PHILIPPART, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (3):
- France (3):
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Centre Hospitalier Bicetre, Paris
  - Hôpital Cochin, Paris

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Prescott HC, Angus DC. Enhancing Recovery From Sepsis: A Review. JAMA. 2018 Jan 2;319(1):62-75. doi: 10.1001/jama.2017.17687. PMID 29297082
- [Background] Brun-Buisson C, Meshaka P, Pinton P, Vallet B; EPISEPSIS Study Group. EPISEPSIS: a reappraisal of the epidemiology and outcome of severe sepsis in French intensive care units. Intensive Care Med. 2004 Apr;30(4):580-8. doi: 10.1007/s00134-003-2121-4. Epub 2004 Mar 2. PMID 14997295
- [Background] Pletz MW, Blasi F, Chalmers JD, Dela Cruz CS, Feldman C, Luna CM, Ramirez JA, Shindo Y, Stolz D, Torres A, Webb B, Welte T, Wunderink R, Aliberti S. International Perspective on the New 2019 American Thoracic Society/Infectious Diseases Society of America Community-Acquired Pneumonia Guideline: A Critical Appraisal by a Global Expert Panel. Chest. 2020 Nov;158(5):1912-1918. doi: 10.1016/j.chest.2020.07.089. Epub 2020 Aug 25. PMID 32858009
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Kumar A. Early antimicrobial therapy in severe sepsis and septic shock. Curr Infect Dis Rep. 2010 Sep;12(5):336-44. doi: 10.1007/s11908-010-0128-x. PMID 21308515
- [Background] Seymour CW, Kahn JM, Martin-Gill C, Callaway CW, Yealy DM, Scales D, Angus DC. Delays From First Medical Contact to Antibiotic Administration for Sepsis. Crit Care Med. 2017 May;45(5):759-765. doi: 10.1097/CCM.0000000000002264. PMID 28234754
- [Background] Whiles BB, Deis AS, Simpson SQ. Increased Time to Initial Antimicrobial Administration Is Associated With Progression to Septic Shock in Severe Sepsis Patients. Crit Care Med. 2017 Apr;45(4):623-629. doi: 10.1097/CCM.0000000000002262. PMID 28169944
- [Background] Skorup P, Maudsdotter L, Lipcsey M, Larsson A, Sjolin J. Mode of bacterial killing affects the inflammatory response and associated organ dysfunctions in a porcine E. coli intensive care sepsis model. Crit Care. 2020 Nov 14;24(1):646. doi: 10.1186/s13054-020-03303-9. PMID 33189146